CLINICAL TRIAL: NCT03155802
Title: Use of Novel Biomarkers and Echocardiography to Assess Subclinical Cardiac Toxicity in Breast Cancer Patients Receiving Anthracyclines
Brief Title: Novel Biomarkers and Echocardiography for Subclinical Cardiac Toxicity in Breast Cancer Patients Receiving Anthracyclines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 922042
Record Dates: First submitted 2017-04-17; First posted 2017-05-16 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Cardiotoxicity; Heart Failure; Breast Cancer; Anthracycline Induced Cardiomyopathy; Biomarkers; Echocardiography
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be kept at -70 degrees of Celsius for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot prospective cohort study, in adult female subjects 18-85 years old with a diagnosis of invasive breast cancer who are planned for anthracycline-inclusive chemotherapy and followed up for a time period of 6 months post completion of anthracycline chemotherapy. They will participate in blood and imaging tests with a goal of determining the best method for predicting the occurrence of cardiotoxicity in this subpopulation.

DETAILED DESCRIPTION:
Anthracyclines and other chemotherapy agents are associated with cardiotoxicity. The risk of cardiac related toxicity is increased in patients with advanced age, with multiple comorbid conditions, and those needing prolonged or intensive treatment. These patients require a tailored approach to surveillance, early diagnosis and treatment of cardiac issues related to cancer therapy, with timely decision making with respect to alterations in therapy. A serum biomarker approach alone or in combination with imaging indices holds promise for early identification, risk stratification and monitoring of chemotherapy related cardiotoxicity.

Thirty-five consecutive adult females between the ages of 18-85 with diagnosis of invasive breast cancer, planned for anthracycline inclusive chemotherapy (+/- taxanes, +/- trastuzumab) will be enrolled.

A detailed medical history (interim where appropriate), physical exam, collection of blood samples for the measurement of Heart Failure (HF) biomarkers (and standard chemistry and hematology parameters), electrocardiogram and a 2D/3D echo cardiogram including the measurement of global longitudinal strain will be performed at baseline, mid chemotherapy, at the end of chemotherapy and 6 months post the completion of chemotherapy. (echocardiogram will not be done during chemotherapy).

The hypothesis being tested in this prospective trial is whether early changes in the levels of serum biomarkers of stress (N terminal pro B-type natriuretic peptide (NT-proBNP)), inflammation (ST2), necrosis (hs troponin), and fibrosis (galectin-3) will correlate with changes in sub-clinical left ventricular dysfunction as assessed by 3-dimensional (3D) echocardiogram with speckle tracking/strain in breast cancer patients receiving anthracycline based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 18-85 years old
2. Biopsy-proven diagnosis of invasive breast cancer carcinoma
3. Plan for anthracycline inclusive chemotherapy (+/- taxanes, +/- trastuzumab)

Exclusion Criteria:

1. History of major heart disease at the time of breast cancer diagnosis (myocardial infarction or known left ventricular dysfunction (LVD) at baseline (defined as ejection fraction <40%)
2. History of known obstructive coronary artery disease (CAD), or coronary revascularization within the past 1 year
3. History of clinical heart failure or previous heart failure hospitalization
4. Patients with elevations in NT-pro BNP (above 3x ULN), or ST2 (above 2x ULN), galectin-3 (above 2x ULN), or hs troponin (above 2x ULN) during baseline screening
5. Patients with metastatic disease or recurrent breast cancer at diagnosis
6. History of other chemotherapy treated malignancy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: females between the ages of 18-85 with diagnosis of invasive breast cancer, planned for anthracycline inclusive chemotherapy (+/- taxanes, +/- trastuzumab).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Association of Heart Failure Biomarkers with Global Longitudinal strain rate | up to 35 weeks
  N Terminal-proBNP, hs troponin, ST2, galectin-3 with global longitudinal strain rate

SECONDARY OUTCOMES:
Prediction of initiation/change in cardiovascular medications based on serum biomarkers | up to 35 weeks
  NT-proBNP
Prediction of initiation/change in cardiovascular medications based on serum biomarkers | up to 35 weeks
  ST2
Prediction of initiation/change in cardiovascular medications based on serum biomarkers | up to 35 weeks
  hs-troponin
Prediction of initiation/change in cardiovascular medications based on serum biomarkers | up to 35 weeks
  galectin-3
Prediction of cardiotoxicity based on serum biomarkers | up to 35 weeks
  galectin-3
Prediction of cardiotoxicity based on serum biomarkers | up to 35 weeks
  NT-proBNP
Prediction of cardiotoxicity based on serum biomarkers | up to 35 weeks
  hs-troponin
Prediction of cardiotoxicity based on serum biomarkers | up to 35 weeks
  ST2

OTHER OUTCOMES:
Association between modifications in chemotherapy with detection of subclinical cardiotoxicity | up to 10 weeks
  frequency of chemotherapy changes with subclinical cardiotoxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No